CLINICAL TRIAL: NCT00861081
Title: RCT of an Intervention to Enable Stroke Survivors in Los Angeles County Hospitals to "Stay Within the Guidelines" (SUSTAIN)
Brief Title: Intervention to Enable Stroke Survivors in Los Angeles County Hospitals to "Stay Within the Guidelines"
Acronym: SUSTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Southern California (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Rancho Los Amigos National Rehabilitation Center (Other); Olive View-UCLA Education & Research Institute (Other); American Heart Association (Other)
Responsible Party: Principal Investigator, Barbara Vickrey, MD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: G-08-07-019-01; 0875133N (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Group Clinics; Self Management
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Care management (Experimental)
  Interventions: Behavioral: Care Management
- 2: Written Materials (Active Comparator)
  Interventions: Behavioral: Written Materials

INTERVENTIONS:
Behavioral: Care Management — Over a period of one year, subjects will participate in two regular stroke clinics, three group clinics, obtain self-management tools, and will receive a series of four scheduled telephone calls by nurse practitioners to review information delivered during the group clinics and help with care coordination. Usual care will also be available.
  Arms: 1: Care management
Behavioral: Written Materials — Educational materials about stroke that will be distributed during the group clinic session will be mailed to these subjects. These materials have been developed by the American Heart Association. Usual care will also be available.
  Arms: 2: Written Materials

SUMMARY:
The purpose of this study is to test a newly developed outpatient care intervention called SUSTAIN (Systematic Use of Stroke Averting Interventions) for improving delivery of stroke preventive services at Los Angeles County hospitals and to measure the costs of running such an intervention.

DETAILED DESCRIPTION:
Patients randomized to SUSTAIN will participate in group clinics about stroke, given self-management tools about stroke, and will be called by nurse practitioners to coordinate their stroke care. Patients randomized to the control arm will be mailed educational materials about stroke. Subjects in either arm are eligible to receive their usual source of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of LAC+USC, Rancho Los Amigos, Olive View-UCLA, or Harbor-UCLA
* Patients who have had an acute transient ischemic attack (TIA) or ischemic stroke or carotid procedure within the last six months
* English or Spanish speaking
* At least 40 years of age
* Capable of giving informed consent (no proxies will be used to obtain consent)
* Blood pressure not optimally controlled (>120/80, at least 72 hours post-stroke)

Exclusion Criteria:

* Age 39 years or younger
* Hemorrhagic stroke
* Patients with severe global disability which would preclude him/her from participating in group clinics
* Patients with advanced dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 months
  Blood pressure at 12 months will be the primary outcome. Blood pressure will also be measured at baseline and at the 3-month mark to track blood pressure during the entire participation period.

SECONDARY OUTCOMES:
Lipid levels | 12 month
  LDL, HDL, triglycerides and total cholesterol will be measured at 12-months. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Medication Adherence | 8 months
  Medication adherence will be measured in a self-report by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Vickrey, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - UCLA, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Background] Cheng EM, Cunningham WE, Towfighi A, Sanossian N, Bryg RJ, Anderson TL, Guterman JJ, Gross-Schulman SG, Beanes S, Jones AS, Liu H, Ettner SL, Saver JL, Vickrey BG. Randomized, controlled trial of an intervention to enable stroke survivors throughout the Los Angeles County safety net to "stay with the guidelines". Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):229-34. doi: 10.1161/CIRCOUTCOMES.110.951012. PMID 21406671
- [Result] Cheng EM, Cunningham WE, Towfighi A, Sanossian N, Bryg RJ, Anderson TL, Barry F, Douglas SM, Hudson L, Ayala-Rivera M, Guterman JJ, Gross-Schulman S, Beanes S, Jones AS, Liu H, Vickrey BG. Efficacy of a Chronic Care-Based Intervention on Secondary Stroke Prevention Among Vulnerable Stroke Survivors: A Randomized Controlled Trial. Circ Cardiovasc Qual Outcomes. 2018 Jan;11(1):e003228. doi: 10.1161/CIRCOUTCOMES.116.003228. PMID 29321134
- [Derived] Richards A, Jackson NJ, Cheng EM, Bryg RJ, Brown A, Towfighi A, Sanossian N, Barry F, Li N, Vickrey BG. Derivation and Application of a Tool to Estimate Benefits From Multiple Therapies That Reduce Recurrent Stroke Risk. Stroke. 2020 May;51(5):1563-1569. doi: 10.1161/STROKEAHA.119.027160. Epub 2020 Mar 23. PMID 32200759